CLINICAL TRIAL: NCT04294732
Title: Efficacy of Popliteal Block and Bupivacaine Concentration Used for Analgesia in Foot and Ankle Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bozyaka Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Hazal Ezgi Çifci, Principal Investigator Hazal Ezgi Çifci, Bozyaka Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HZLEZGCFCANLEKR
Record Dates: First submitted 2018-09-27; First posted 2020-03-04 (Actual); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: Foot and Ankle Surgery; Popliteal Nerve Block; Peripheral Nerve Block
MeSH Terms: interventions — Bupivacaine; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: The study was designed to be prospective and randomized. Patients will be divided into 3 groups by simple randomization. The results of power analysis (G-power 3.1) revealed that a total of 60 patients were required to be included in the study. Because of that approximately 20 patients are planned for each group
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Spinal anesthesia will be performed in all three groups. During procedure 8 ml saline with 8 ml bupivacaine will be apply to the first group and 8 ml bupivacaine and 16 ml of saline will be apply to the second group. Only spinal anesthesia will be given to the third group without peripheral nerve block. The patients participating in the study will not be informed about which group they belong to, the person who makes the block will not prepare the drug and the person who makes the block, the patient and the nurse will not know which concentration drug applied to which patient.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Only spinal anesthesia (Placebo Comparator): Only spinal anesthesia without peripheral nerve block
  Interventions: Drug: Only spinal anesthesia without peripheral nerve block
- high concentration (Active Comparator): 8 ml saline with 8 ml bupivacaine
  Interventions: Drug: Bupivacaine
- low concentration (Experimental): 8 ml bupivacaine with 16 ml of saline
  Interventions: Drug: Bupivacaine

INTERVENTIONS:
Drug: Bupivacaine — bupivacaine is a local anesthetic drug which is already using in surgical procedures.
  saline is isotonic solution of which has include %0,9 NACL.
  Other Names: Saline
  Arms: high concentration; low concentration
Drug: Only spinal anesthesia without peripheral nerve block — Only spinal anesthesia without peripheral nerve block
  Arms: Only spinal anesthesia

SUMMARY:
In the orthopedic foot and ankle surgeries, the effects of postoperative popliteal nerve block applied for palliation of pain and local anesthetic agent in two different concentrations (0.166 and 0.250) which were used in popliteal nerve block procedure, will be investigated.

DETAILED DESCRIPTION:
USG guided popliteal nerve block known to be effective in postoperative pain management in foot and ankle surgical procedures but clinical use of the procedure is not yet widespread. However, the volume and concentration of local anesthetic drugs to be administered is still controversial. The study was designed to be prospective and randomized. Patients will be divided into 3 groups by simple randomization. The results of power analysis (G-power 3.1) revealed that a total of 60 patients were required to be included in the study. Because of that, approximately 20 patients are planned for each group. Spinal anesthesia will be performed in all three groups. During procedure 8 ml saline with 8 ml bupivacaine will be apply to the first group and 8 ml bupivacaine and 16 ml of saline will be apply to the second group. Only spinal anesthesia will be given to the third group without peripheral nerve block. The patients participating in the study will not be informed about which group they belong to, the person who makes the block will not prepare the drug and the person who makes the block, the patient and the nurse will not know which concentration drug applied to which patient. Between two groups duration of motor block, duration of sensory block, post-op analgesia time, mobilization time will be investigate. Also the first pain time, the opioid requirement and opioid dose used will be investigated. Analgesia, duration of analgesia, time and requirement of administered IV analgesics, mobilization time after popliteal nerve block will be investigate. package statistical program SPSS (Statistical Package for Social Sciences version 18) will be used for statistical analysis. The parametrical values from the descriptive values will be given as mean and standard deviation, the non-parametric values will be given as number and percentage or median and min-max value. The suitability of the data to the normal distribution will be evaluated with the Kolmogorov-Smirnov test. One-way ANOVA will be use for the comparison of the quantitative data which is appropriate to the normal distribution. The Tukey HSD test will be used to identify the group that caused the difference. Kruskal Wallis-H test will be used to compare quantitative parameters that do not show normal distribution. Mann Whitney U test will be applied to determine the cause of the difference and chi-square test will be used to compare qualitative data. For the analyzes, the level of significance in the 95% confidence interval was found in p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients undergoing orthopedic surgery on foot and ankle and who agreed to participate in the study

Exclusion Criteria:

* Patients with sensitivity to local anesthetic
* Patients who do not want to be included in the study
* Preoperative mobilization and movement limitation
* Patients who are not co-operate, cannot complete questionnaire forms and inquiry forms
* Patients with skin infection at the injection site
* Patients with diabetic neuropathy
* Patients with bleeding disorder / Coagulopathy
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
pain relief activity of popliteal nerve block within thirty-six hours | Postoperative 12th hour
  Numeric rating scale will be use for evaluate pain. Numeric rating scale contains 0 to 10 pain scores. 0 means no pain and 10 means maximum pain perception which is described by patient. Numeric rating scale will be apply to patient at 12th hour. İf the numeric rating scale is above 3, it will be considered as pain.
pain relief activity of popliteal nerve block within thirty-six hours | Postoperative 24th hour
  Numeric rating scale will be use for evaluate pain. Numeric rating scale contains 0 to 10 pain scores. 0 means no pain and 10 means maximum pain perception which is described by patient. Numeric rating scale will be apply to patient at 24th hour. İf the numeric rating scale is above 3, it will be considered as pain.
pain relief activity of popliteal nerve block within thirty-six hours | Postoperative 36th hour
  Numeric rating scale will be use for evaluate pain. Numeric rating scale contains 0 to 10 pain scores. 0 means no pain and 10 means maximum pain perception which is described by patient. Numeric rating scale will be apply to patient at 36th hour. İf the numeric rating scale is above 3, it will be considered as pain.
pain relief activity of popliteal nerve block within three months | Postoperative first month
  Numeric rating scale will be use for evaluate pain. Numeric rating scale contains 0 to 10 pain scores. 0 means no pain and 10 means maximum pain perception which is described by patient. Numeric rating scale will be apply to patient at first months. İf the numeric rating scale is above 3, it will be considered as pain.
pain relief activity of popliteal nerve block within three months | Postoperative second month
  Numeric rating scale will be use for evaluate pain. Numeric rating scale contains 0 to 10 pain scores. 0 means no pain and 10 means maximum pain perception which is described by patient. Numeric rating scale will be apply to patient at second months. İf the numeric rating scale is above 3, it will be considered as pain. İf pain persist over 1 month, ıt will be considered as chronic pain.
pain relief activity of popliteal nerve block within three months | Postoperative third month
  Numeric rating scale will be use for evaluate pain. Numeric rating scale contains 0 to 10 pain scores. 0 means no pain and 10 means maximum pain perception which is described by patient. Numeric rating scale will be apply to patient at third months. İf the numeric rating scale is above 3, it will be considered as pain. İf pain persist over 1 month, ıt will be considered as chronic pain.

SECONDARY OUTCOMES:
Investigate the pain relief activity of different concentrations within thirty-six hours | Postoperative 12th hour.
  To compare the pain relief activity of bupivacaine at a concentration of 0.166 and 0.250 in popliteal block. Numeric rating scale will be use for evaluate pain Numeric rating scale contains 0 to 10 pain scores. 0 means no pain and 10 means maximum pain perception which is described by patient. Numeric rating scale will be apply to patient at 12th hour. İf the numeric rating scale is above 3, it will be considered as pain.
Investigate the pain relief activity of different concentrations within thirty-six hours | Postoperative 24th hour
  To compare the pain relief activity of bupivacaine at a concentration of 0.166 and 0.250 in popliteal block. Numeric rating scale will be use for evaluate pain Numeric rating scale contains 0 to 10 pain scores. 0 means no pain and 10 means maximum pain perception which is described by patient. Numeric rating scale will be apply to patient at 24th hours. İf the numeric rating scale is above 3, it will be considered as pain.
Investigate the pain relief activity of different concentrations within thirty-six hours | Postoperative 36th hour
  To compare the pain relief activity of bupivacaine at a concentration of 0.166 and 0.250 in popliteal block. Numeric rating scale will be use for evaluate pain Numeric rating scale contains 0 to 10 pain scores. 0 means no pain and 10 means maximum pain perception which is described by patient. Numeric rating scale will be apply to patient at 36th hours. İf the numeric rating scale is above 3, it will be considered as pain.
Investigate the pain relief activity of different concentrations within three months | Postoperative first month
  To compare the pain relief activity of bupivacaine at a concentration of 0.166 and 0.250 in popliteal block. Numeric rating scale will be use for evaluate pain Numeric rating scale contains 0 to 10 pain scores. 0 means no pain and 10 means maximum pain perception which is described by patient. Numeric rating scale will be apply to patient at first month. İf the numeric rating scale is above 3, it will be considered as pain.
Investigate the pain relief activity of different concentrations within three months | Postoperative second month
  To compare the pain relief activity of bupivacaine at a concentration of 0.166 and 0.250 in popliteal block. Numeric rating scale will be use for evaluate pain Numeric rating scale contains 0 to 10 pain scores. 0 means no pain and 10 means maximum pain perception which is described by patient. Numeric rating scale will be apply to patient at second month. İf the numeric rating scale is above 3, it will be considered as pain. İf pain persist over 1 month, ıt will be considered as chronic pain.
Investigate the pain relief activity of different concentrations within three months | Postoperative third month
  To compare the pain relief activity of bupivacaine at a concentration of 0.166 and 0.250 in popliteal block. Numeric rating scale will be use for evaluate pain Numeric rating scale contains 0 to 10 pain scores. 0 means no pain and 10 means maximum pain perception which is described by patient. Numeric rating scale will be apply to patient at third month. İf the numeric rating scale is above 3, it will be considered as pain. İf pain persist over 1 month, ıt will be considered as chronic pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Hazal Ezgi Çifci, Izmir, Eyalet/Yerleşke, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided